CLINICAL TRIAL: NCT01759186
Title: Severe Asthma Research Program
Brief Title: Airway Redox and Gender Determinants in Severe Asthma
Acronym: SARP3
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Case Western Reserve University (Other); University of Virginia (Other)
Responsible Party: Principal Investigator, Serpil Erzurum, multiple Prinicipal Investigators [B Gaston, S. Erzurum, G. Teague], The Cleveland Clinic
Other Study IDs: 6185
Record Dates: First submitted 2012-11-16; First posted 2013-01-03 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Asthma
Keywords: Asthma; Biomakers; Phenotype
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- None interventional

SUMMARY:
The investigators will study the biologic and chemical differences that cause the greater incidence, and severity of asthma in women as compared to men. Severe asthma affects boys more than girls, while severe asthma in adults is predominantly a disease of women. The investigators aim to identify the processes that occur in the body that are behind the onset of severe asthma in young women during the teenage years, and the resolution of severe asthma in boys. To further evaluate gender influences on asthma, asthmatic women at different stages of their menstrual cycle (period) will be also studied. The investigators aim to use biomarkers to develop testing procedures that will identify different types or characteristics of asthma in men and women; and to follow patients over time to uncover relevant clinical outcomes of biomarkers. The investigators anticipate that they will 1) develop clinically relevant tests to identify unique types or characteristics of asthma and severe asthma; 2) determine outcomes over time of biochemically-defined types of asthma; and 3) identify the reasons for why adult women are affected more than men with severe asthma.

DETAILED DESCRIPTION:
This scientific site-specific project is part of a larger network of asthma studies, the Severe Asthma Research Program (SARP). The mission of SARP is to improve the understanding of severe asthma to develop better treatments.

ELIGIBILITY:
Inclusion Criteria:

Subjects with asthma

* children age 6-17 years old (25% enrollment)
* adults 18 years and older (75% enrollment)

Exclusion Criteria:

* Pregnancy during the characterization phase
* Current smoking
* Smoking history > 10 pack years if ≥30 years of age, or smoking history > 5 pack years if <30 years of age (Note: if a subject has a smoking history, no smoking within the past year),
* Other chronic pulmonary disorders associated with asthma-like symptoms, including (but not limited to) cystic fibrosis, chronic obstructive pulmonary disease, chronic bronchitis, vocal cord dysfunction (that is the sole cause of respiratory symptoms and at the PI's discretion)
* Severe scoliosis or chest wall deformities
* History of premature birth before 35 weeks gestation
* Unwillingness to receive an intramuscular triamcinolone acetonide injection.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients living in the greater Cleveland area, and in Virginia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-12; Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Identify metabolic mechanism(s) and age dependent change in the epidemiology of asthma | 5 years
  To determine if asthma severity is worsened in females with changes in estradiol that occur during puberty as measured by asthma control tests and lung functions

SECONDARY OUTCOMES:
Development of clinical testing procedures to assign metabolic asthma phenotypes | 5 years
  To determine if urine and blood and exhaled metabolic biomarkers can predict asthma phenotypes and severity as measured by lung functions and asthma control tests

OTHER OUTCOMES:
Gender influences on severe asthma | 5 years
  To determine if adult women have more severe asthma in relation to menstrual cycle as measured by lung functions and remodeling on biopsies of the airway.

CONTACTS AND LOCATIONS:
Overall Officials: Serpil C Erzurum, MD, Principal Investigator — The Cleveland Clinic; Benjamin Gaston, MD, Principal Investigator — Case Western Reserve University; W. Gerald Teague, MD, Principal Investigator — University of Virginia
Locations (4):
- United States (4):
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Dunican EM, Elicker BM, Gierada DS, Nagle SK, Schiebler ML, Newell JD, Raymond WW, Lachowicz-Scroggins ME, Di Maio S, Hoffman EA, Castro M, Fain SB, Jarjour NN, Israel E, Levy BD, Erzurum SC, Wenzel SE, Meyers DA, Bleecker ER, Phillips BR, Mauger DT, Gordon ED, Woodruff PG, Peters MC, Fahy JV; National Heart Lung and Blood Institute (NHLBI) Severe Asthma Research Program (SARP). Mucus plugs in patients with asthma linked to eosinophilia and airflow obstruction. J Clin Invest. 2018 Mar 1;128(3):997-1009. doi: 10.1172/JCI95693. Epub 2018 Feb 5. PMID 29400693